CLINICAL TRIAL: NCT02778594
Title: Pharmacokinetic-pharmacodynamic Interaction Between Three Different Single Doses of BIA 3-202 and a Single-dose of Controlled-release 100/25 mg Levodopa/Benserazide (Madopar® HBS 125): a Double-blind, Randomised, Four-way Crossover, Placebo-controlled Study in Healthy Volunteers
Brief Title: Pharmacokinetic-pharmacodynamic Interaction Between BIA 3-202 and Levodopa/Benserazide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-3202-108
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Parkinson's Disease (PD)
MeSH Terms: conditions — Parkinson Disease | interventions — nebicapone; Levodopa; Benserazide; benserazide, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo (4 tablets) Simultaneously with the placebo dose, subjects were administered 1 capsule of Madopar® HBS 125
  Interventions: Drug: Placebo; Drug: levodopa 100 mg / benserazide 25 mg
- Nebicapone 50 mg (Experimental): Nebicapone 50 mg (1 tablet of 50 mg plus 3 tablets of placebo). Simultaneously with the nebicapone dose, subjects were administered 1 capsule of Madopar® HBS 125
  Interventions: Drug: BIA 3-202; Drug: Placebo; Drug: levodopa 100 mg / benserazide 25 mg
- Nebicapone 100 mg (Experimental): Nebicapone 100 mg (2 tablets of 50 mg plus 2 tablets of placebo). Simultaneously with the nebicapone dose, subjects were administered 1 capsule of Madopar® HBS 125
  Interventions: Drug: BIA 3-202; Drug: Placebo; Drug: levodopa 100 mg / benserazide 25 mg
- Nebicapone 200 mg (Experimental): Nebicapone 200 mg (4 tablets of 50 mg). Simultaneously with the nebicapone dose, subjects were administered 1 capsule of Madopar® HBS 125
  Interventions: Drug: BIA 3-202; Drug: levodopa 100 mg / benserazide 25 mg

INTERVENTIONS:
Drug: BIA 3-202 — nebicapone 50 mg tablets; oral use
  Other Names: Nebicapone
  Arms: Nebicapone 100 mg; Nebicapone 200 mg; Nebicapone 50 mg
Drug: Placebo — Nebicapone matching placebo tablets
  Arms: Nebicapone 100 mg; Nebicapone 50 mg; Placebo
Drug: levodopa 100 mg / benserazide 25 mg — Madopar® HBS 125 (levodopa 100 mg / benserazide 25 mg) capsules; oral use
  Other Names: Madopar

SUMMARY:
The purpose of this study is to determine the effect of three single oral doses of nebicapone (50 mg, 100 mg and 200 mg) on the levodopa pharmacokinetics when administered in combination with a single-dose of controlled release levodopa 100 mg/benserazide 25 mg (Madopar® HBS 125).

DETAILED DESCRIPTION:
STUDY DESIGN AND METHODOLOGY:

Single centre, double-blind, randomised, placebo-controlled, 4-way crossover study with 4 single-dose treatment periods. The washout period between doses was 5 days or more.

Screening: Subjects were screened for eligibility within 28 and 7 days before first admission. The screening consisted of: medical history; physical examination, vital signs; complete neurological examination; 12-lead ECG; haematology, coagulation, plasma biochemistry and urinalysis tests; HIV, hepatitis B and hepatitis C serology; drugs of abuse and alcohol screen; urine pregnancy test in women of childbearing potential; and review of the selection criteria.

Treatment periods: In each treatment period, eligible subjects were admitted to the UFH on the day prior to receiving the study medication for: vital signs; medical history and physical examination updates; 12-lead ECG; haematology and plasma biochemistry; drugs of abuse and alcohol screen; and urine pregnancy test in women of childbearing potential. On first admission, subjects had a review of the selection criteria and were randomly assigned to one of the treatment sequences. On the morning of the dosing day, subjects received a dose of nebicapone/placebo concomitantly with a dose of Madopar® HBS 125 in fasting conditions (at least 8 hours) and remained in the UFH until at least 24 h post-dose; then, they left and returned for the next period or the follow-up visit. At given time-points between pre-dose and discharge, subjects were submitted to vital signs recording, brief neurological examination, 12-lead ECG, and blood sampling for plasma drug determination and erythrocyte S-COMT activity assay. At discharge, vital signs and ECG were recorded, and haematology and plasma biochemistry tests were performed. Blood samples (7 mL) for the determination of plasma concentration of levodopa, 3-O-methyldopa (3-OMD) and nebicapone, and for the assay of the erythrocyte S-COMT activity were taken at the following times: pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose.

Follow-up: A follow-up visit occurred approximately 7-10 days after discharge of last treatment period or early discontinuation for: medical history and physical examination updates; vital signs; 12-lead ECG; haematology, plasma biochemistry and urinalysis tests; and pregnancy test in women of childbearing potential.

ELIGIBILITY:
Inclusion Criteria:

Subjects were eligible for entry into the study if they fulfilled the following inclusion criteria:

* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Subjects who had clinical laboratory test results clinically acceptable at screening and admission to first treatment period.
* Subjects who had negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening.
* Subjects who had a negative screen for alcohol and drugs of abuse at screening and admission to each treatment period.
* Subjects who were non-smokers or who smoked ≤ 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier, intrauterine device or abstinence.
* (If female) She had a negative urine pregnancy test at screening and admission to each treatment period.

Exclusion Criteria:

Subjects were not eligible for entry into the study if they fulfilled the following exclusion criteria:

* Subjects who did not conform to the above inclusion criteria, or
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of glaucoma.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 21 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening or first admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening or first admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had used medicines within 2 weeks of first admission that, in the opinion of the investigator, may affect the safety or other study assessments.
* Subjects who had used any investigational drug or participated in any clinical trial within 2 months of their first admission.
* Subjects who had donated or received any blood or blood products within the previous 2 months prior to screening.
* Subjects who were vegetarians, vegans or have medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not use an approved effective contraceptive method (double-barrier, intra-uterine device or abstinence) or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2005-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) | pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose
  Mean Cmax pharmacokinetic parameters of levodopa following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or nebicapone
Time of occurrence of Cmax (tmax) | pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose
  Mean tmax pharmacokinetic parameters of levodopa following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or nebicapone
Area under the plasma concentration-time curve (AUC) from time zero to the last sampling time at which concentrations were at or above the limit of quantification (AUC0-t) | pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose
  Mean AUC0-t pharmacokinetic parameters of levodopa following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or nebicapone
Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞) | pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose
  Mean AUC0-00 pharmacokinetic parameters of levodopa following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or nebicapone
Apparent terminal half-life, calculated from ln 2/λz (t1/2) | pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 h post-dose
  Mean t1/2 pharmacokinetic parameters of levodopa following oral administration of single-doses of Madopar® HBS 125 concomitantly with placebo or nebicapone

CONTACTS AND LOCATIONS:
Locations (1):
- Human Pharmacology Unit, S. Mamede Do Coronado, Portugal

IPD SHARING:
Plan to Share IPD: Undecided